CLINICAL TRIAL: NCT03543670
Title: Efficacy of Oncoxin-Viusin® Nutritional Supplement Related With the Onco-specific Treatments in Prostate Cancer Patients
Brief Title: Evaluation of Oncoxin-Viusid® in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-4
Record Dates: First submitted 2018-05-03; First posted 2018-06-01 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncoxin-Viusid (Experimental)
  Interventions: Dietary Supplement: Oncoxin-Viusid

INTERVENTIONS:
Dietary Supplement: Oncoxin-Viusid — Support treatment with Oncoxin-Viusid (75mL/day) during chemotherapy/Radiotherapy until two weeks after (a total of 8 months).

SUMMARY:
A not randomized clinical survey was done in 25 pacients with histological diagnosis confirmed of a prostatic adenocarcinoma and hardy in hormonotherapy at the Calixto Garcia Hospital in Habana (2016-2018).

Researches had as identifying goal the efecctiveness study of Oncoxin-Viusid® nutritional supplement as a support to convencional treatment. The patient were treated with habitual doses of Docetacel and 75 mg per day of supplement during and fiften day after the quimiotherapy. The rest of numbers and severety of adverse reactions were determined as well as its influences on life quality when this co-therapy is performed, the evaluation of progresion spare survival and the porcentage of recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Masculine >18 years-old patients
* Performans status: Karnofsky ≥ 70 or (ECOG <2)
* Hormonal treatment alternatives 6 or 8 weeks before the inclusion ,with resistence to hormonal treatments
* Normal laboratory tests to onco-specific treatments.
* Ecocardiogram with a eyección fraction > 60 %, in patients with history of cardiovascular deseases.
* Patients with life expectative more than 6 months.

Exclusion Criteria:

* Patients who are receiving another onco-specific product in research.
* Patients with known hypersensitivity to anthracyclines and / or mitoxantrone
* Decompensated intercurrent diseases, including: active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, liver damage and psychiatric illnesses that could limit adherence to the requirements of the clinical trial or any other special condition that at the discretion of the physician put your health and life at risk during the study or your participation in the trial.
* Patients with cerebral metastases.
* Patients with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 12 months
  General quality of life (EORTC QLQ C30 questionnaire and specific for prostate cancer EORTC QLQ - PR25)
Adverse events | 12 months
  Toxicity (hematological, hemochemistry, clinical response) stablished by WHO

SECONDARY OUTCOMES:
Overal survival | 12 months
  Global Survival Rate (GSR)
Overal recurrences | 12 months
  Progression-free survival - PFS

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes I. Fundora, Dr., Principal Investigator — General Calixto García University Hospital
Locations (1):
- General Calixto García University Hospital, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Fundora Ramos MI, Maden LB, Casanova FO, Cruz FH, Reyes CS, Gato AH, Lyncon IB, Gonzalez EV, Morales KP, Lence JJ, Sanz E. Oncoxin-Viusid(R) may improve quality of life and survival in patients with hormone-refractory prostate cancer undergoing onco-specific treatments. Mol Clin Oncol. 2021 Jan;14(1):5. doi: 10.3892/mco.2020.2167. Epub 2020 Nov 5. PMID 33235733